CLINICAL TRIAL: NCT00861900
Title: Immune Mechanisms of Rejection in Human Lung Allografts
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 98-0977-201103312; HL056643
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators have obtained compelling evidence that the development of anti-human leukocyte antigen (anti-HLA) antibodies against mismatched donor antigens significantly correlates with the development of bronchiolitis obliterans (BOS). Further, these anti-HLA antibodies are developed at least 15 months prior to any clinical evidence of BOS. This lag period between the development of anti-HLA antibodies and the onset of BOS gives us an opportunity to intervene to delay and/or prevent the development of BOS.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipient.

Exclusion Criteria:

* Pregnant women,
* Prisoners, AND
* Anyone who is unable or unwilling to consent to this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who is a candidate for a lung transplant.
Sampling Method: Non-Probability Sample
Enrollment: 778 (Actual)
Dates: Start 1998-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy event is the change in pulmonary function testing values (FEV1). | Lung function is monitored at regular intervals. Patients will be followed for five years.

SECONDARY OUTCOMES:
Secondary efficacy measurements include allograft and patient survival, incidence of BOS and Obliterative bronchiolitis. | The subjects are monitored at regular intervals. Patients will be followed for five years.

CONTACTS AND LOCATIONS:
Overall Officials: Thalachallour Mohanakumar, PhD, Principal Investigator — Washington University School of Medicine